CLINICAL TRIAL: NCT04228445
Title: An Open-Label Study of Two Different Doses of 3,3'-Dioxo-2,2'-Bisindolylidene-5,5'-Disulfonate Disodium 0.8% Solution When Used as an Aid for Ureteral Patency
Brief Title: 3,3'-Dioxo-2,2'-Bisindolylidene-5,5'-Disulfonate Disodium 0.8% Solution as an Aid for Ureteral Patency
Acronym: UP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Prove pharm (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: PVP-19IC01
Record Dates: First submitted 2019-12-23; First posted 2020-01-14 (Actual); Results first posted 2022-11-30 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Ureter Injury

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- HIGH DOSE (Experimental): 48 subjects randomly treated with 5 mL of drug
  Interventions: Drug: 3,3'-Dioxo-2,2'-bisindolylidene-5,5'-disulfonate disodium 0.8%; Drug: Saline spray
- LOW DOSE (Experimental): 48 subjects randomly treated with 2.5 mL of drug
  Interventions: Drug: 3,3'-Dioxo-2,2'-bisindolylidene-5,5'-disulfonate disodium 0.8%; Drug: Saline spray
- Saline (Placebo Comparator): 96 subjects treated with 5 ml of saline than crossover to treatment arm
  Interventions: Drug: Saline spray

INTERVENTIONS:
Drug: 3,3'-Dioxo-2,2'-bisindolylidene-5,5'-disulfonate disodium 0.8% — Experimental contrast dye that is commonly used as a visualization aid in pelvic and abdominal surgeries and for various diagnostic procedures in medical practice.
  Arms: HIGH DOSE; LOW DOSE
Drug: Saline spray — Placebo

SUMMARY:
To determine whether the use of 3,3'-Dioxo-2,2'-Bisindolylidene-5,5'-Disulfonate Disodium 0.8% Solution for injection provides a visualization advantage compared to saline when used as an aid in the determination of ureteral patency

DETAILED DESCRIPTION:
This is an open-label, randomized, multicenter study to evaluate the efficacy, safety, and pharmacokinetics of two doses (2.5 mL and 5.0 mL) of 3,3'-Dioxo-2,2'-bisindolylidene-5,5'-disulfonate disodium solution for injection when used as an aid in the determination of ureteral patency. Study will enroll up to 116 subjects from approximately 10 study centers in the United States.

ELIGIBILITY:
Inclusion Criteria:

* Subjects between ≥ 18 and ≤ 85 years old.
* Subjects who signed written, IRB approved, informed consent form.
* Subjects scheduled for urological or gynecological surgical procedures in which the patency of the ureter must be assessed by the surgeon during the procedure

Exclusion Criteria:

* Subjects with stage 4 or 5 Chronic Kidney Failure as evidenced by a GFR <30 mL/min/1.73m2 (using the MDRD) or need for dialysis in the near future, or having only 1 kidney.
* Subjects with known severe hypersensitivity reactions to IC or other dyes including contrast agents.
* Known history of drug or alcohol abuse within 6 months prior to the time of screening visit.
* Subjects, as assessed by the Investigator, with conditions/concomitant diseases precluding their safe participation in this study (e.g. major systemic diseases).
* Unable to meet specific protocol requirements (e.g., scheduled visits) or subject is uncooperative or has a condition that could lead to non-compliance with the study procedures.
* Subject is the Investigator or any Sub-Investigator, research assistant, pharmacist, study coordinator, other staff or relative thereof directly involved in the conduct of the protocol;
* Subjects with life expectancy < 6 months;
* Requirement for concomitant treatment that could bias primary evaluation.
* Subjects who are pregnant or breast-feeding.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2020-02-13 (Actual); Primary Completion 2021-06-03 (Actual); Study Completion 2021-06-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Todd Koch, Study Director — Prove pharm
Locations (1):
- Adult and Pediatric Urology, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a crossover study where each subject served as their own control, so each subject received the control (saline solution) was evaluated for the endpoints and then received either the high or low dose based on their randomization assignment. So the total number of participants were 121 although each participant provided data for one of the active groups and the saline group.
Groups:
- SALINE Then HIGH DOSE: Approximately 48 subjects treated with 5 ml of saline than crossover to be treated with 5 mL of drug
  3,3'-Dioxo-2,2'-bisindolylidene-5,5'-disulfonate disodium 0.8%: Experimental contrast dye that is commonly used as a visualization aid in pelvic and abdominal surgeries and for various diagnostic procedures in medical practice.
  Saline solution: Placebo
- SALINE Then LOW DOSE: Approximately 48 subjects treated with 5 ml of saline than crossover to be treated with 2.5 mL of drug
  3,3'-Dioxo-2,2'-bisindolylidene-5,5'-disulfonate disodium 0.8%: Experimental contrast dye that is commonly used as a visualization aid in pelvic and abdominal surgeries and for various diagnostic procedures in medical practice.
  Saline solution: Placebo
Period: Overall Study
Arm/Group | SALINE Then HIGH DOSE | SALINE Then LOW DOSE
Started | 62 | 59
Completed | 59 | 55
Not Completed | 3 | 4
Not completed — Lost to Follow-up | 1 | 1
Not completed — Physician Decision | 1 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Planned procedure not performed after randomization, study drug not administered | 1 | 0

BASELINE CHARACTERISTICS:
Population: Population presented is the Safety Analysis Set, while the population presented in the Participant Flow was the all randomized population
Groups:
- Total: Total of all reporting groups
Arm/Group | SALINE Then HIGH DOSE | SALINE Then LOW DOSE | Total
Number analyzed (Participants) | 60 | 58 | 118
Age, Customized [Count of Participants; unit: Participants]
  < 65 years old | 42 | 41 | 83
  >/= 65 years to <75 years old | 11 | 12 | 23
  >/= 75 years old | 7 | 5 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 45 | 87
  Male | 18 | 13 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 8 | 18
  Not Hispanic or Latino | 50 | 48 | 98
  Unknown or Not Reported | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 4 | 8
  White | 56 | 49 | 105
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 3 | 3
Region of Enrollment [Number; unit: participants]
  United States | 60 | 58 | 118

OUTCOME MEASURES:

1. Primary Outcome: Urine Jet Conspicuity Score
Description: The urine jet conspicuity score provided by the blinded central review process as assessed by the following 5-point ordinal scale.
  1. = No jet observed
  2. = Weak jet, little color contrast
  3. = Color contrast or significant jet flow
  4. = Strong jet flow with good color contrast
  5. = Strong jet flow with striking contrast in color
Time Frame: 10 minutes
Population: The efficacy analysis set, also referred to as the modified intent-to-treat (mITT) analysis set, included all subjects in the safety analysis set who had a surgical procedure to assess ureteral patency, who received both study drugs (saline and indigo carmine), and a video approximately 10 minutes in length was available after each treatment.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- HIGH DOSE: Approximately 48 subjects randomly treated with 5 mL of drug
  3,3'-Dioxo-2,2'-bisindolylidene-5,5'-disulfonate disodium 0.8%: Experimental contrast dye that is commonly used as a visualization aid in pelvic and abdominal surgeries and for various diagnostic procedures in medical practice.
  Saline solution: Placebo
- LOW DOSE: Approximately 48 subjects randomly treated with 2.5 mL of drug
  3,3'-Dioxo-2,2'-bisindolylidene-5,5'-disulfonate disodium 0.8%: Experimental contrast dye that is commonly used as a visualization aid in pelvic and abdominal surgeries and for various diagnostic procedures in medical practice.
  Saline solution: Placebo
- Saline: Approximately 96 subjects treated with 5 ml of saline than crossover to treatment arm
  Saline solution: Placebo
Arm/Group | HIGH DOSE | LOW DOSE | Saline
Number analyzed (Participants) | 49 | 47 | 96
score on a scale | 4.1 (1.34) | 4.2 (1.17) | 2.5 (1.10)
Statistical Analysis 1: Comparison: HIGH DOSE vs Saline; Test type: Superiority; p < 0.0001, Score statistics for Type 3 GEE analysis; Odds Ratio (OR) = 14.041, 95% CI 2-sided [7.394 to 26.662]
Statistical Analysis 2: Comparison: LOW DOSE vs Saline; Test type: Superiority; p < 0.0001, Score statistics for Type 3 GEE analysis; Odds Ratio (OR) = 16.772, 95% CI 2-sided [8.625 to 32.617]

2. Secondary Outcome: Percentage of Responders
Description: A subject was a responder when there was ≥1-point improvement in the urine jet conspicuity scores following the indigo carmine versus saline treatment (indigo carmine - saline ≥1) and the conspicuity score following the indigo carmine treatment was 3, 4, or 5. The responder criteria were assessed separately for each ureter for each subject based on the blinded central reviewer's conspicuity score.
Time Frame: 10 Minutes
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | HIGH DOSE | LOW DOSE
Number analyzed (Participants) | 49 | 47
Participants
  Responder | 43 | 41
  Non-Responder | 6 | 6
Statistical Analysis 1: Comparison: HIGH DOSE; Test type: Other; Percentage of Responders = 87.8, 95% CI 2-sided [78.6 to 96.9] — Missing data imputed as non-responder
Statistical Analysis 2: Comparison: LOW DOSE; Test type: Other; Percentage of Responders = 87.2, 95% CI 2-sided [77.7 to 96.8] — Missing data imputed as non-responder

3. Secondary Outcome: Physician Satisfaction Agreement Scale
Description: After the completion of the procedure, the surgeon rated the experience of using indigo carmine for each subject using the 5-point PSAS, in which:
  "Compared to the use of saline treatment, my ability to assess ureteral patency was improved after the addition of indigo carmine."
  1. = Strongly Agree
  2. = Agree
  3. = Neither Agree nor Disagree
  4. = Disagree
  5. = Strongly Disagree
  The surgeon was considered satisfied with the indigo carmine treatment if his/her rating was either a 1 (strongly agree) or a 2 (agree); otherwise, the surgeon was considered unsatisfied with the indigo carmine treatment.
Time Frame: 10 Minutes
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | HIGH DOSE | LOW DOSE
Number analyzed (Participants) | 49 | 47
Participants
  Satisfied (score of 1 or 2) | 44 | 38
  Unsatisfied (Score of 3,4 or 5) | 5 | 9
Statistical Analysis 1: Comparison: HIGH DOSE; Test type: Other; percentage of satisfaction = 89.8, 95% CI 2-sided [78.2 to 95.6]
Statistical Analysis 2: Comparison: LOW DOSE; Test type: Other; percentage of satisfaction = 80.9, 95% CI 2-sided [67.5 to 89.6]

4. Secondary Outcome: Time to Visualization
Description: Time to visualization (minutes) of blue color in the ureteral jets flow following indigo carmine treatment
Time Frame: 10 Minutes
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Minutes
Arm/Group | HIGH DOSE | LOW DOSE
Number analyzed (Participants) | 49 | 47
Minutes | 6.00 [5.25 to 7.00] | 5.93 [5.12 to 7.00]
Statistical Analysis 1: Comparison: HIGH DOSE; Test type: Other; median time to visualization (minutes) = 6.00, 95% CI 2-sided [5.25 to 7.00]
Statistical Analysis 2: Comparison: LOW DOSE; Test type: Other; median time to visualization (minutes) = 5.93, 95% CI 2-sided [5.12 to 7.00]

5. Other Pre Specified Outcome: Surgeon Urine Jet Conspicuity Score
Description: The urine jet conspicuity score provided by the surgeon as assessed by the following 5-point ordinal scale.
  1. = No jet observed
  2. = Weak jet, little color contrast
  3. = Color contrast or significant jet flow
  4. = Strong jet flow with good color contrast
  5. = Strong jet flow with striking contrast in color
Time Frame: 10 Minutes
Population: The efficacy analysis set, also referred to as the modified intent-to-treat (mITT) analysis set, included all subjects in the safety analysis set who had a surgical procedure to assess ureteral patency, who received both study drugs (saline and indigo carmine), and a video approximately 10 minutes in length was available after each treatment (subjects with missing data excluded).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HIGH DOSE | LOW DOSE | Saline
Number analyzed (Participants) | 47 | 46 | 93
score on a scale | 4.2 (1.31) | 4.2 (1.26) | 2.4 (1.07)
Statistical Analysis 1: Comparison: HIGH DOSE vs Saline; Test type: Superiority; p < 0.0001, Score statistics for Type 3 GEE analysis; Odds Ratio (OR) = 19.532, 95% CI 2-sided [8.738 to 43.663]
Statistical Analysis 2: Comparison: LOW DOSE vs Saline; Test type: Superiority; p < 0.0001, Score statistics for Type 3 GEE analysis; Odds Ratio (OR) = 15.730, 95% CI 2-sided [7.199 to 34.369]

6. Other Pre Specified Outcome: Concordance of Conspicuity Scores
Description: Concordance of conspicuity scores between the surgeons' assessments and the blinded central reviewer assessments. If the difference between raters in conspicuity score was within ±1 (ie, the difference ranged from 1 to +1, inclusive), the scores were considered to agree.
  The urine jet conspicuity score as assessed by the following 5-point ordinal scale.
  1. = No jet observed
  2. = Weak jet, little color contrast
  3. = Color contrast or significant jet flow
  4. = Strong jet flow with good color contrast
  5. = Strong jet flow with striking contrast in color
Time Frame: 10 Min
Population: mITT Analysis Set; Subjects Without Missing Surgeon or Central Assessment Data
Measure: Count of Participants; unit: Participants
Arm/Group | HIGH DOSE | LOW DOSE | Saline
Number analyzed (Participants) | 45 | 43 | 88
Participants
  Left Ureter: Agreement | 41 | 38 | 67
  Left Ureter: Disagreement | 4 | 5 | 21
  Right ureter: Agreement | 43 | 37 | 63
  Right ureter: Disagreement | 2 | 6 | 25
Statistical Analysis 1: Comparison: HIGH DOSE; Left Ureter; Test type: Other; Percentage of Agreement = 91.1
Statistical Analysis 2: Comparison: LOW DOSE; Left Ureter; Test type: Other; Percentage of Agreement = 88.4
Statistical Analysis 3: Comparison: Saline; Left Ureter; Test type: Other; Percentage of Agreement = 76.1
Statistical Analysis 4: Comparison: HIGH DOSE; Right Ureter; Test type: Other; Percentage of Agreement = 95.6
Statistical Analysis 5: Comparison: LOW DOSE; Right Ureter; Test type: Other; Percentage of Agreement = 86.0
Statistical Analysis 6: Comparison: Saline; Right Ureter; Test type: Other; Percentage of Agreement = 71.6

7. Other Pre Specified Outcome: Conspicuity Score Difference Between the Indigo Carmine High Dose and Indigo Carmine Low Dose by Central Review Process
Description: Exploratory analysis of the urine jet conspicuity score difference between the indigo carmine high dose and indigo carmine low dose by central review Process
  The urine jet conspicuity score provided by the blinded central review process as assessed by the following 5-point ordinal scale.
  1. = No jet observed
  2. = Weak jet, little color contrast
  3. = Color contrast or significant jet flow
  4. = Strong jet flow with good color contrast
  5. = Strong jet flow with striking contrast in color
Time Frame: 10 minutes
Population: mITT Analysis Set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HIGH DOSE | LOW DOSE
Number analyzed (Participants) | 49 | 47
score on a scale | 4.1 (1.34) | 4.2 (1.17)
Statistical Analysis 1: Comparison: HIGH DOSE vs LOW DOSE; Test type: Superiority; p = 0.4595, Score statistics for Type 3 GEE analysis; Odds Ratio (OR) = 0.771, 95% CI 2-sided [.388 to 1.534]

8. Other Pre Specified Outcome: Conspicuity Score Difference Between the Indigo Carmine High Dose and Indigo Carmine Low Dose as Assessed by Surgeons Who Were Blinded to the Dose of Indigo Carmine
Description: Exploratory analysis of conspicuity score difference between the indigo carmine high dose and indigo carmine low dose as assessed by surgeons who were blinded to the dose of indigo carmine
  The urine jet conspicuity score as assessed by the following 5-point ordinal scale.
  1. = No jet observed
  2. = Weak jet, little color contrast
  3. = Color contrast or significant jet flow
  4. = Strong jet flow with good color contrast
  5. = Strong jet flow with striking contrast in color
Time Frame: 10 Minutes
Population: mITT population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HIGH DOSE | LOW DOSE
Number analyzed (Participants) | 47 | 46
score on a scale | 4.2 (1.31) | 4.2 (1.26)
Statistical Analysis 1: Comparison: HIGH DOSE vs LOW DOSE; Test type: Superiority; p = 0.9220, Score statistics for Type 3 GEE analysis; Odds Ratio (OR) = 1.036, 95% CI 2-sided [.509 to 2.110]

ADVERSE EVENTS:
Time Frame: Saline group: AEs collected from the time of saline administration until the beginning of indigo carmine administration (approximately 10 minutes) IC groups AEs collected from the start of IC administration until 30 (+/- 2) days post surgery
Description: AEs were collected through non leading questioning of participants as well as via scheduled post treatment evaluation of clinical laboratories, physical exam, vital signs and EKGs.
Arm/Group | HIGH DOSE | LOW DOSE | Saline
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/58 | 0/118
Serious Adverse Events (participants affected / at risk) | 1/60 | 3/58 | 0/118
Other Adverse Events (participants affected / at risk) | 14/60 | 14/58 | 0/118
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HIGH DOSE (N=60) | LOW DOSE (N=58) | Saline (N=118)
Pneumonia aspiration (Aspiration pneumonia) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Bilateral PE) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Left iliac DVT) (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1.7% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HIGH DOSE (N=60) | LOW DOSE (N=58) | Saline (N=118)
Constipation (Gastrointestinal disorders) | 3 (3) | 3 (3) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 4 (4) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (7):
  • Study Protocol: Original protocol (2019-07-01): https://cdn.clinicaltrials.gov/large-docs/45/NCT04228445/Prot_000.pdf
  • Study Protocol: Administrative change #1 (2019-10-18): https://cdn.clinicaltrials.gov/large-docs/45/NCT04228445/Prot_001.pdf
  • Study Protocol: Amendment #1 (2019-12-10): https://cdn.clinicaltrials.gov/large-docs/45/NCT04228445/Prot_002.pdf
  • Study Protocol: Clarification Letter #1 (2020-06-23): https://cdn.clinicaltrials.gov/large-docs/45/NCT04228445/Prot_003.pdf
  • Study Protocol: Amendment #2 (2020-09-02): https://cdn.clinicaltrials.gov/large-docs/45/NCT04228445/Prot_004.pdf
  • Study Protocol: Clarification Letter #2 (2020-12-18): https://cdn.clinicaltrials.gov/large-docs/45/NCT04228445/Prot_005.pdf
  • Statistical Analysis Plan (2021-06-26): https://cdn.clinicaltrials.gov/large-docs/45/NCT04228445/SAP_006.pdf